CLINICAL TRIAL: NCT04829487
Title: The Role of Vitamin D Supplementation on Pain in Women With Primary Dysmenorrhea and Hypovitaminosis D: A Randomized, Double-blind, Placebo-Controlled Study
Brief Title: The Role of Vitamin D Supplementation on Pain in Women With Primary Dysmenorrhea and Hypovitaminosis D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Preeyaporn Jirakittidul, Doctor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 247/2021
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Vitamin D 50,000 IU orally weekly for 8 weeks
  Interventions: Drug: Ergocalciferol Capsules
- Placebo (Placebo Comparator): Placebo capsules orally weekly for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol Capsules — Given to subjects 50,000 IU per week for 8 weeks
  Other Names: Vitamin D2
  Arms: Vitamin D
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of vitamin D supplementation on the pain score of primary dysmenorrhea. Our hypothesis is that by normalizing vitamin D level could help improve pain score of women who have primary dysmenorrhea.

DETAILED DESCRIPTION:
This study is aimed to be conducted in randomised controlled trial, comparing between intervention group and placebo group. We include women with primary dysmenorrhea who also have low vitamin D level in this trial. Our primary outcome is to compare visual analog pain scale between intervention and placebo group after treatment. After randomised and allocated, these women will be given vitamin D 50,000 IU or placebo capsules orally weekly for 8 consecutive weeks. We monitor pain score daily from the cycle before the drugs started until complete 8-week course of the regimen mentioned. Also vitamin D levels will be monitored twice, one before treatment and the other after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhea
* Hypovitaminosis D

Exclusion Criteria:

* Using calcium, magnesium or phosphorus in the past 3 months
* Using hormonal contraception or IUD in the past 6 months
* No smoking or alcohol drinking
* Chronic underlying diseases
* Allergic to components in study drugs

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog pain scale | 8 weeks
  Pain score between intervention and placebo group after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mananya Silpakit, Doctor, Principal Investigator — Reproductive medicine unit, Department of OB-GYN, Faculty of Medicine, Siriraj Hospital

IPD SHARING:
Plan to Share IPD: No